CLINICAL TRIAL: NCT05034770
Title: Effectiveness of Major Ozone Autohemotherapy in the Treatment of Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Emine Dundar Ahi, MD (Other)
Responsible Party: Sponsor-Investigator, Emine Dundar Ahi, MD, Principal Investigator, Kocaeli University
Organization: Kocaeli University (Other)
Other Study IDs: 2020-161
Record Dates: First submitted 2021-05-21; First posted 2021-09-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: major ozone autohemotherapy — This treatment is based on treating 100 ml of the pa- tient's blood with 100 ml of O3 followed by reinfusion in the donor, in a fast procedure. Each patient received 10 sessions of autohemotherapy with O3 twice a week.

SUMMARY:
Patients who were admitted to the Physical Medicine and Rehabilitation (PMR) outpatient clinic of our hospital between January 2017 and December 2020 and were treated with Major ozone autohemotherapy with a diagnosis of Fibromyalgia syndrome will include to the study. Visual anolog scale (VAS), Fibromyalgia Impact Questionnare (FIQ) and Short Form Health Survey-36 (SF-36) scores of the patients before and after treatment were recorded. Statistical analysis of these outcome scores will be made.

ELIGIBILITY:
Exclusion Criteria:

* has pregnancy,
* has primary romatological disease,
* has primary psychiatric disease
* <18, >60 years old patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * 18-60 years ranged, male and female patients
  * diagnosed fibromyalgia syndrome witc ACR 1990,2010 criterias,
  * volunteers that gave consent,
  * treated with major ozone autohemotherapy (10 sessions)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Short Form Health Survey-36 | 20 minutes
  the 36-item Short Form Health Survey (SF-36) is a measure of health-related quality-of-life. It allows assessment across eight health domains: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). The scores of these eight domains can also be summated in two major categories: physical composite score (PCS) and mental composite score (MCS) to reflect the overall physical and mental health, respectively. Scores of 100 for PF, RP, BP, SF, and RE domains and scores of 50 in the remaining three domains, GH, VT, and MH, indicate an absence of problems in those areas.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnare | 5 minutes
  The Fibromyalgia Impact Questionnare (FIQ) is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. It has been designed to measure the components of health status that are believed to be most affected by FM. FIQ is scored in such a way that a higher score indicates a greater impact of the syndrome on the person. Each of the 10 items has a maximum possible score of 10. Thus the maximum possible score is 100. The average FM patient scores about 50, severely afflicted patients are usually 70 plus.

OTHER OUTCOMES:
Visual Analog Scale (VAS) | 10 seconds
  The Visual Analog Scale (VAS) is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. FM patients mark the point on the line that best corresponds to their symptom severity. To this end, they are instructed to put a cross on the straight line at the point that most accurately expresses their degree of agreement. When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. If documented in paper form, the scores can then be simply transferred to a 100-value scale using a millimeter tape measure. The division into hundredths is considered sufﬁciently sensitive.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Medar Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No